CLINICAL TRIAL: NCT03545022
Title: Acupuncture on Anxiety and Inflammatory Events Following Surgery of Mandibular Third Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of the Valleys of Jequitinhonha and Mucuri (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1.688.806
Record Dates: First submitted 2018-05-04; First posted 2018-06-04 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Tooth Extraction; Molar, Third; Pain, Postoperative; Trismus; Edema; Anxiety
Keywords: third molar; acupuncture; pain; edema; trismus; anxiety
MeSH Terms: conditions — Pain, Postoperative; Trismus; Edema; Anxiety Disorders; Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients who met the study criteria were randomized to the type of acupuncture (active acupuncture or placebo acupuncture) and to the side of the first surgery (right or left). The randomization was performed by a researcher not involved in the study by lottery. Four papers in two opaque envelopes were used, one with the side of the teeth and another with the protocol of acupuncture treatment to be received, protocol 1 or 2.
  The patients, the surgeon, the acupuncturist and the investigator were unaware of which acupuncture treatment was used at each surgery (active or placebo). In order to conceal the randomization, the needles for the active and placebo protocol were identical and were delivered to the acupuncturist in two boxes labeled protocol 1 and 2 and the codes were revealed only after completion of the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active acupuncture (Active Comparator): For both types of treatment, 0.25x30mm stainless steel needles were used (Dux, Brazil).The protocols were differentiated by needle size, in which the placebo needle is not inserted into the patient's skin and has an identical appearance to the active needle.The needle measuring 0.25x30mm was used as an active needle. The needles were inserted partially into an opaque guide tube filled with condensation silicone. This process was used to simulate the needle insertion for the patient and the acupuncturist and for the needle support. The active needle as well as the placebo needle were attached to the skin with an adhesive pedestal to hold the needle in place, even without inserting it into the skin.
  Interventions: Procedure: Acupuncture
- Placebo acupuncture (Placebo Comparator): For both types of treatment, 0.25x30mm stainless steel needles were used (Dux, Brazil).The protocols were differentiated by needle size, in which the placebo needle is not inserted into the patient's skin and has an identical appearance to the active needle. In the placebo needle, the needles were cut in 5mm, to measure 0.25x25mm. The needles were inserted partially into an opaque guide tube filled with condensation silicone. This process was used to simulate the needle insertion for the patient and the acupuncturist and for the needle support. The active needle, as well as the placebo needle, were attached to the skin with an adhesive pedestal to hold the needle in place, even without inserting it into the skin.
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — The application of acupuncture was performed in four sessions, 30 minutes prior to surgery, 24, 48 and 72 hours following the surgery, before variables measurements. The points were manually stimulated and the needles were inserted up to 4mm. There were 11 points, applied bilaterally, two of them, point VG20 and Yintang, for anxiety control, only at the preoperative time and not bilateral. The points to reduce pain, edema, and trismus were IG4 (Hegu), F3 (Taichong) and E44 (Neiting), TA21 (Ermen), ID19 (Ting-Kong), E6 (Jiagle) and E7 (Towei) , point B60 (Kunlum) and VB34 (Yanglingquan). All patients received the same treatment in all sessions.
  After the needle devices were inserted, the needles were re-stimulated manually once after 10 minutes and removed after more 10 minutes.

SUMMARY:
The aim of this study was to compare the effect of acupuncture and placebo acupuncture for the control of pain, edema, and trismus following the extraction of third molars and control of preoperative anxiety. Patients who met the study criteria were randomized to the type of acupuncture (active acupuncture or placebo acupuncture) and to the side of the first surgery (right or left).

DETAILED DESCRIPTION:
Studies using acupuncture have shown promising results in the control of pain, edema, trismus and anxiety control. The use of this technique is interesting considering the negative effects of excessive use of medicines and the side effects of medications which are the most common treatment used for the control of these complications. However, there are no reports in the literature that evaluated the effects of acupuncture on the control of these variables following mandibular third molar extraction, using the placebo-needle design and blinding the patients, operators, and evaluators. Therefore, the aim of this split-mouth randomized triple-blind clinical trial was to compare the efficacy of acupuncture and placebo acupuncture for the control of pain, edema, trismus and preoperative anxiety in the extraction of third molars.

ELIGIBILITY:
Inclusion Criteria:

* Patients with indication for bilateral extraction of asymptomatic mandibular third molars in the position class IIB, according to the classification of Pell & Gregory (1933).

Exclusion Criteria:

* Previous use of any type of medication in the 15 days prior to the study;
* Hypersensitivity to drugs, substances or any materials used in this experiment;
* Pregnancy or lactation;
* Previous case of pericoronitis;
* People who have previously undergone any kind of acupuncture treatment.

Ages: 17 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Presence and intensity of postoperative pain at 24 hours following the surgery | The marking was performed at 24 hours postoperatively.
  For the evaluation of the presence and intensity of postoperative pain, a coded record (Protocol 1 or 2) was used, identifying the patient, the operated side and the chronology of the intervention (first or second surgery). Each record contained three visual analog scales (VAS) with a 10 cm line, without demarcations, with the number 0 (no pain) on the left edge and the number 10 on the right edge (extreme pain). The volunteers were instructed to mark, with a vertical trace, the point of the scale that best defined their degree of painful sensitivity after surgical procedures, which was measured with a ruler afterward.
Presence and intensity of postoperative pain at 48 hours following the surgery. | The marking was performed at 48 hours postoperatively.
  For the evaluation of the presence and intensity of postoperative pain, a coded record (Protocol 1 or 2) was used, identifying the patient, the operated side and the chronology of the intervention (first or second surgery). Each record contained three visual analog scales (VAS) with a 10 cm line, without demarcations, with the number 0 (no pain) on the left edge and the number 10 on the right edge (extreme pain). The volunteers were instructed to mark, with a vertical trace, the point of the scale that best defined their degree of painful sensitivity after surgical procedures, which was measured with a ruler afterward.
Presence and intensity of postoperative pain at 72 hours following the surgery. | The marking was performed at 72 hours postoperatively.
  For the evaluation of the presence and intensity of postoperative pain, a coded record (Protocol 1 or 2) was used, identifying the patient, the operated side and the chronology of the intervention (first or second surgery). Each record contained three visual analog scales (VAS) with a 10 cm line, without demarcations, with the number 0 (no pain) on the left edge and the number 10 on the right edge (extreme pain). The volunteers were instructed to mark, with a vertical trace, the point of the scale that best defined their degree of painful sensitivity after surgical procedures, which was measured with a ruler afterward.
Change from baseline facial swelling (edema) at 24 hours following the surgery. | The measurements were obtained preoperatively (baseline) and at 24 hours following the surgery.
  Facial swelling (edema) was determined by measuring with tape measure according to the method described by Gabka and Matsumara (1971). Three measurements were performed between the 5 reference points: tragus, pogonium (soft tissues), lateral corner of the eyes, the angle of the mandible, external corner of the mouth. The sum of the preoperative measurements was the standard of normality for each side. The swelling evaluation was done by subtracting the postoperative measurements by the sum obtained at the preoperative moment (baseline).
Change from baseline facial swelling (edema) at 48 hours following the surgery. | The measurements were obtained preoperatively (baseline) and at 48 hours following the surgery.
  Facial swelling (edema) was determined by measuring with tape measure according to the method described by Gabka and Matsumara (1971). Three measurements were performed between the 5 reference points: tragus, pogonium (soft tissues), lateral corner of the eyes, the angle of the mandible, external corner of the mouth. The sum of the preoperative measurements was the standard of normality for each side. The swelling evaluation was done by subtracting the postoperative measurements by the sum obtained at the preoperative moment (baseline).
Change from baseline facial swelling (edema) at 72 hours following the surgery. | The measurements were obtained preoperatively (baseline) and at 72 hours following the surgery.
  Facial swelling (edema) was determined by measuring with tape measure according to the method described by Gabka and Matsumara (1971). Three measurements were performed between the 5 reference points: tragus, pogonium (soft tissues), lateral corner of the eyes, the angle of the mandible, external corner of the mouth. The sum of the preoperative measurements was the standard of normality for each side. The swelling evaluation was done by subtracting the postoperative measurements by the sum obtained at the preoperative moment (baseline).
Change from baseline facial swelling (edema) at 7 days following the surgery. | The measurements were obtained preoperatively (baseline) and at 7 days following the surgery.
  Facial swelling (edema) was determined by measuring with tape measure according to the method described by Gabka and Matsumara (1971). Three measurements were performed between the 5 reference points: tragus, pogonium (soft tissues), lateral corner of the eyes, the angle of the mandible, external corner of the mouth. The sum of the preoperative measurements was the standard of normality for each side. The swelling evaluation was done by subtracting the postoperative measurements by the sum obtained at the preoperative moment (baseline).
Change from baseline mouth opening at 24 hours following the surgery. | The measurement was determined in the preoperative period (baseline) and at the period of 24 hours following the surgery.
  The maximum mouth opening was used to assess the level of trismus. The distance between the left upper and lower incisor was measured with a digital caliper and transcribed, in millimeters, for data recording. After verification of the measurements in the postoperative period, the difference in the measurements before and after the surgical procedure was observed, determining the level of trismus.
Change from baseline mouth opening at 48 hours following the surgery. | The measurement was determined in the preoperative period (baseline) and at the period of 48 hours following the surgery.
  The maximum mouth opening was used to assess the level of trismus. The distance between the left upper and lower incisor was measured with a digital caliper and transcribed, in millimeters, for data recording. After verification of the measurements in the postoperative period, the difference in the measurements before and after the surgical procedure was observed, determining the level of trismus.
Change from baseline mouth opening at 72 hours following the surgery. | The measurement was determined in the preoperative period (baseline) and at the period of 72 hours following the surgery.
  The maximum mouth opening was used to assess the level of trismus. The distance between the left upper and lower incisor was measured with a digital caliper and transcribed, in millimeters, for data recording. After verification of the measurements in the postoperative period, the difference in the measurements before and after the surgical procedure was observed, determining the level of trismus.
Change from baseline mouth opening at 7 days following the surgery. | The measurement was determined in the preoperative period (baseline) and at the period of 7 days following the surgery.
  The maximum mouth opening was used to assess the level of trismus. The distance between the left upper and lower incisor was measured with a digital caliper and transcribed, in millimeters, for data recording. After verification of the measurements in the postoperative period, the difference in the measurements before and after the surgical procedure was observed, determining the level of trismus.
Change of anxiety state scores using STAI questionnaire at the moment before the preoperative acupuncture and after the acupuncture. | The STAI-S questionnaires were applied before the preoperative acupuncture and after acupuncture.
  Anxiety was evaluated with the Spielberger State-Trait Anxiety Inventory (STAI) questionnaire, translated and validated to Portuguese by Biaggio et al. (1977). The STAI is a validated questionnaire consisting of two parts, each with 20 questions. One part, STAI-S, evaluates the state of anxiety which is defined as anxiety in response to a situation. The other part, STAI-T, evaluates the anxiety trait, defined by the level of anxiety normally felt by the person. The two parts can be scored from 20 to 80, with the highest values indicating the highest rates of anxiety. Values ≥40 indicate a high level of anxiety and ≥50 as very high.
Change of anxiety state scores using a Visual Analogue Scale (VAS) questionnaire at the moment before the preoperative acupuncture and after the acupuncture. | The VAS were applied before the preoperative acupuncture and after acupuncture.
  A visual analog scale (VAS) consisted of a 10cm line, without divisions was used. The patients were instructed to mark the level of anxiety at that moment, with the "0" without anxiety and "10", with a high level of anxiety, that was measured with a ruler later.

SECONDARY OUTCOMES:
Duration of surgery | From the time of the initial incision to the time of the final suture.
  The duration of surgery was recorded with a stopwatch in seconds.
Number of painkillers tablets | By the seventh postoperative day.
  The number of paracetamol tablets taken after the surgery was registered by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Catharina V Armond, Principal Investigator — Federal University of Jequitinhonha and Mucuri Valleys

IPD SHARING:
Plan to Share IPD: No